CLINICAL TRIAL: NCT02344407
Title: Partnership for Research on Ebola Vaccines in Liberia (PREVAIL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 999915071; 15-I-N071 (Other: NIH IRB Protocol ID number)
Record Dates: First submitted 2015-01-22; First posted 2015-01-26 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Ebola Virus
Keywords: Zaire Ebola Virus Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Experimental): ChAd3-EBO Z
  Interventions: Biological: ChAd3-EBO Z
- 3 (Experimental): VSVG-ZEBOV
  Interventions: Biological: VSVG-ZEBOV
- 1 (Placebo Comparator): Placebo (Saline)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VSVG-ZEBOV — The VSVdeltaG-ZEBOV vaccine is comprised of a single recombinant (vesicular stomatitis virus) VSV isolate (11481 nt) modified to replace the gene encoding the G envelope glycoprotein with the gene encoding the envelope glycoprotein from the Ebola virus Zaire strain (ZEBOV)
  Arms: 3
Biological: ChAd3-EBO Z — The ChAd3-EBO Z vaccine is comprised of a ChAd3 vector with a DNA fragment insert that encodes the Ebola virus glycoprotein, which is expressed on the virion surface and is critical for attachment to host cells and catalysis of membrane fusion.
  Arms: 2
Biological: Placebo
  Arms: 1

SUMMARY:
Background:

- Ebola virus disease (EVD) affects many people in Liberia and other countries in West Africa. It is caused by the Ebola virus and makes people sick with fever, headache, vomiting, diarrhea, rash, and bleeding. About half the people with EVD die. There is no approved treatment for it. Researchers are studying two Ebola vaccines. The vaccines do not cause Ebola.

Objectives:

- To study the safety and efficacy of two Ebola vaccines.

Eligibility:

- Adults 18 and older who live in Liberia and are at risk for Ebola infection but have never had Ebola.

Design:

* Participants will give information including birthdate, gender, occupation, and location of home. They will give contact information for themselves and 2 alternate contacts. They will give a history of their contact with people with Ebola. Some participants may have a physical. They may have blood taken.
* Participants will be injected with either an Ebola vaccine or a placebo with a needle in the upper arm. The placebo is a salt solution.
* Participants will have blood taken.
* Participants will be watched for 30 minutes.
* Participants will return to the clinic 1 week and 1 month after they get the shot. They will have blood taken.
* After that, participants will be contacted monthly to discuss how they are feeling. They may be contacted by phone, may visit the clinic, or may have a home visit.
* The study ends 8-12 months after participants get the shot. If one of the vaccines works against Ebola and does not have many side effects, participants can get the vaccine if they did not get it in the study.

DETAILED DESCRIPTION:
Ebola virus disease (EVD) in West Africa is spreading rapidly, and there is a critical need for a vaccine to prevent EVD. There are two candidate Ebola virus vaccines, the chimpanzee adenovirus 3 (ChAd3-EBO Z)-based vaccine and the Vesicular Stomatitis virus (VSVdeltaG-ZEBOV)-based vaccine. This study will evaluate both of these vaccines in a randomized, double-blind, controlled, 3-arm study in Liberia. Each vaccine will be compared against the same active control. Because there are limited data on the safety of these vaccines, the initial phase (phase 2) of the study will include the collection of more detailed data on safety and will define the immune response elicited by each vaccine in the first 600 volunteers. With the decline in new cases of Ebola virus infection the phase 3 component was no longer deemed to be feasible and, following safety, ethical and FDA approve/concurrence, the study was amended to a more robust, 1,500 person phase 2 design.

With the amendment to only a phasae 3 study the endpoint reverted to the phase 2 endpoint of safety and immunogenicity.

Participants aged 18 year and older will be enrolled at health clinics in Monrovia, Liberia over 4 months. A single dose of the assigned agent will be administered. Participants in phase 2 will undergo blood draw and assessment of adverse events (AEs) and signs and symptoms of Ebola infection at 1 week and 1 month after vaccination, and monthly assessment of AEs and signs and symptoms of Ebola thereafter. Participants in phase 3 will undergo monthly assessment of AEs and signs and symptoms of Ebola infection after vaccination. All participants will be followed for 8 to 12 months.

This clinical trial to evaluate vaccine efficacy will provide an accurate assessment of the benefits and risks associated with each candidate vaccine and inform policy on wider scale vaccination in other countries.

ELIGIBILITY:
* INCLUSION CRITERIA:

The inclusion criteria for the study are broad reflecting the target population that would eventually receive an efficacious vaccine.

* Informed consent
* Age greater than or equal to 18 years
* Likely to be in the surrounding area of the vaccination center for at least one year.

EXCLUSION CRITERIA:

* Fever greater than or equal to 38.0 degrees Celsius
* History of EVD (self-report)
* Current pregnancy (a negative urine pregnancy test is required for women of child-bearing potential)
* Breast-feeding an infant
* Any condition which would limit the ability of the participant to meet the requirements of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2015-01-20; Primary Completion 2016-06-01 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Clifford Lane, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Liberian Ministry of Health and Social Welfare, Monrovia, Liberia

REFERENCES:
- [Background] Feldmann H, Geisbert TW. Ebola haemorrhagic fever. Lancet. 2011 Mar 5;377(9768):849-62. doi: 10.1016/S0140-6736(10)60667-8. PMID 21084112
- [Background] Chertow DS, Kleine C, Edwards JK, Scaini R, Giuliani R, Sprecher A. Ebola virus disease in West Africa--clinical manifestations and management. N Engl J Med. 2014 Nov 27;371(22):2054-7. doi: 10.1056/NEJMp1413084. Epub 2014 Nov 5. No abstract available. PMID 25372854
- [Background] Colloca S, Barnes E, Folgori A, Ammendola V, Capone S, Cirillo A, Siani L, Naddeo M, Grazioli F, Esposito ML, Ambrosio M, Sparacino A, Bartiromo M, Meola A, Smith K, Kurioka A, O'Hara GA, Ewer KJ, Anagnostou N, Bliss C, Hill AV, Traboni C, Klenerman P, Cortese R, Nicosia A. Vaccine vectors derived from a large collection of simian adenoviruses induce potent cellular immunity across multiple species. Sci Transl Med. 2012 Jan 4;4(115):115ra2. doi: 10.1126/scitranslmed.3002925. PMID 22218691
- [Derived] Simon JK, Kennedy SB, Mahon BE, Dubey SA, Grant-Klein RJ, Liu K, Hartzel J, Coller BG, Welebob C, Hanson ME, Grais RF. Immunogenicity of rVSVDeltaG-ZEBOV-GP Ebola vaccine (ERVEBO(R)) in African clinical trial participants by age, sex, and baseline GP-ELISA titer: A post hoc analysis of three Phase 2/3 trials. Vaccine. 2022 Nov 2;40(46):6599-6606. doi: 10.1016/j.vaccine.2022.09.037. Epub 2022 Oct 5. PMID 36208978
- [Derived] Antonello J, Grant-Klein RJ, Nichols R, Kennedy SB, Dubey S, Simon JK. Serostatus cutoff levels and fold increase to define seroresponse to recombinant vesicular stomatitis virus - Zaire Ebola virus envelope glycoprotein vaccine: An evidence-based analysis. Vaccine. 2020 Jun 26;38(31):4885-4891. doi: 10.1016/j.vaccine.2020.04.061. Epub 2020 Jun 1. PMID 32499064
- [Derived] Logue J, Tuznik K, Follmann D, Grandits G, Marchand J, Reilly C, Sarro YDS, Pettitt J, Stavale EJ, Fallah M, Olinger GG, Bolay FK, Hensley LE. Use of the Filovirus Animal Non-Clinical Group (FANG) Ebola virus immuno-assay requires fewer study participants to power a study than the Alpha Diagnostic International assay. J Virol Methods. 2018 May;255:84-90. doi: 10.1016/j.jviromet.2018.02.018. Epub 2018 Feb 23. PMID 29481881
- [Derived] Kennedy SB, Bolay F, Kieh M, Grandits G, Badio M, Ballou R, Eckes R, Feinberg M, Follmann D, Grund B, Gupta S, Hensley L, Higgs E, Janosko K, Johnson M, Kateh F, Logue J, Marchand J, Monath T, Nason M, Nyenswah T, Roman F, Stavale E, Wolfson J, Neaton JD, Lane HC; PREVAIL I Study Group. Phase 2 Placebo-Controlled Trial of Two Vaccines to Prevent Ebola in Liberia. N Engl J Med. 2017 Oct 12;377(15):1438-1447. doi: 10.1056/NEJMoa1614067. PMID 29020589
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166

RESULTS

PARTICIPANT FLOW:
Groups:
- ChAd3-EBO Z: ChAd3-EBO Z
  ChAd3-EBO Z: The ChAd3-EBO Z vaccine is comprised of a ChAd3 vector with a DNA fragment insert that encodes the Ebola virus glycoprotein, which is expressed on the virion surface and is critical for attachment to host cells and catalysis of membrane fusion.
- VSVG-ZEBOV: VSVG-ZEBOV
  VSVG-ZEBOV: The VSVdeltaG-ZEBOV vaccine is comprised of a single recombinant (vesicular stomatitis virus) VSV isolate (11481 nt) modified to replace the gene encoding the G envelope glycoprotein with the gene encoding the envelope glycoprotein from the Ebola virus Zaire strain (ZEBOV)
- Placebo (Saline): Placebo
Period: Overall Study
Arm/Group | ChAd3-EBO Z | VSVG-ZEBOV | Placebo (Saline)
Started | 500 | 500 | 500
Completed | 492 | 491 | 494
Not Completed | 8 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ChAd3-EBO Z | VSVG-ZEBOV | Placebo (Saline) | Total
Number analyzed (Participants) | 500 | 500 | 500 | 1500
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [25 to 38] | 29 [24 to 36] | 30 [24 to 39] | 30 [24 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 187 | 177 | 549
  Male | 315 | 313 | 323 | 951
Region of Enrollment [Number; unit: participants]
  Liberia | 500 | 500 | 500 | 1500
Contact past month with someone who had Ebola [Count of Participants; unit: Participants] | 1 | 5 | 5 | 11
Work involves contact with persons with Ebola [Count of Participants; unit: Participants] | 22 | 25 | 22 | 69
HIV Positive [Count of Participants; unit: Participants] | 25 | 22 | 31 | 78
Syphilis positive [Count of Participants; unit: Participants] | 30 | 22 | 25 | 77
IgG antibody level (EU/mL) [Median (Inter-Quartile Range); unit: EU/mL] | 75 [44 to 135] | 81 [49 to 141] | 79 [50 to 148] | 78 [47 to 139]
Positive antibody response [Count of Participants; unit: Participants] | 16 | 18 | 26 | 60

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events.
Description: Number of Participants Experiencing Serious Adverse Events in First 30 Days
Time Frame: One month
Population: All Participants Randomized
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO Z | VSVG-ZEBOV | Placebo (Saline)
Number analyzed (Participants) | 500 | 500 | 500
Participants | 6 | 6 | 8
Statistical Analysis 1: Comparison: ChAd3-EBO Z vs Placebo (Saline); Each active vaccine is compared to the placebo group; Test type: Superiority; p = 0.68, Chi-squared; Bernards Exact Test Chi-square
Statistical Analysis 2: Comparison: VSVG-ZEBOV vs Placebo (Saline); Test type: Superiority; p = 0.68, Chi-squared; Barnard Exact Test Chi-square

2. Primary Outcome: Immunogenicity Measures (ELISA and Neutralization Antigen-specific Assays for Antibody.
Description: Antibody Response at 1-Month (EU/mL) for Participants Without Elevated Levels at Entry
Time Frame: One month
Population: Participants with 1-month antibody data without elevated antibody levels at entry
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | ChAd3-EBO Z | VSVG-ZEBOV | Placebo (Saline)
Number analyzed (Participants) | 478 | 477 | 471
EU/mL | 621 [565 to 682] | 1000 [910 to 1099] | 75 [69 to 80]
Statistical Analysis 1: Comparison: ChAd3-EBO Z vs Placebo (Saline); Test type: Superiority; p < 0.001, ANCOVA; Linear regression (analysis of covariance) adjusted for baseline antibody level
Statistical Analysis 2: Comparison: VSVG-ZEBOV vs Placebo (Saline); Test type: Superiority; p < 0.001, ANCOVA; Analysis of covariance adjusting for baseline antibody level

ADVERSE EVENTS:
Time Frame: First 30 days after vaccination
Arm/Group | ChAd3-EBO Z | VSVG-ZEBOV | Placebo (Saline)
All-Cause Mortality (participants affected / at risk) | 0/500 | 0/500 | 1/500
Serious Adverse Events (participants affected / at risk) | 6/500 | 6/500 | 8/500
Other Adverse Events (participants affected / at risk) | 0/500 | 0/500 | 0/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChAd3-EBO Z (N=500) | VSVG-ZEBOV (N=500) | Placebo (Saline) (N=500)
Malaria (Infections and infestations) | 2 (2) | 6 (6) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pheumocystis jirovecii pheumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No